CLINICAL TRIAL: NCT02138162
Title: A Phase 1, Non-randomized, Open-label, Single-dose Study to Investigate the Pharmacokinetics, Safety and Tolerability of Enzalutamide in Male Subjects With Severe Hepatic Impairment and Normal Hepatic Function
Brief Title: A Study to Investigate the Effect of Severely Diminished Liver Function on the Metabolism, Safety, and Tolerability of a Single Oral Dose of Enzalutamide in Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 9785-CL-0404; 2012-004858-29 (EudraCT Number)
Record Dates: First submitted 2014-05-12; First posted 2014-05-14 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Severe Hepatic Impairment; Normal Hepatic Function
Keywords: Phase 1; Pharmacokinetics; Safety; Severe hepatic impairment; Enzalutamide
MeSH Terms: interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1:Single dose of enzalutamide in hepatically impaired subjects (Experimental): Single dose of enzalutamide
  Interventions: Drug: enzalutamide
- 2:Single dose of enzalutamide in healthy subjects (Experimental): Single dose of enzalutamide
  Interventions: Drug: enzalutamide

INTERVENTIONS:
Drug: enzalutamide — oral
  Other Names: ASP9785,; MDV3100,; Xtandi

SUMMARY:
The influence of severely diminished liver function on the metabolism, safety, and tolerability of a single oral dose of enzalutamide in a group of 8 men. The results are compared to the data gained from 8 age- and BMI-matched men with normal liver function.

DETAILED DESCRIPTION:
Screening takes place between Day -22 and Day -2, and subjects are admitted to the clinic on Day -1. Each subject receives a single oral dose of enzalutamide on Day 1, under fasted conditions. They are discharged on Day 7; ambulant visits take place until Day 50. An End of Study Visit (ESV) occurs 7-10 days after the last PK sampling or early withdrawal.

Full PK profiles are obtained for enzalutamide, metabolite 1 of enzalutamide (M1) and metabolite 2 of enzalutamide (M2) up to 1176 hours (Day 50) after administration.

Safety assessments are performed throughout the study. For subjects with severe hepatic impairment, additional Child-Pugh classification and laboratory safety tests (including liver function tests) are performed regularly after administration.

ELIGIBILITY:
Inclusion Criteria:

* Male subject and their female spouse/partners who are of childbearing potential must be using highly effective contraception consisting of two forms of birth control starting at Screening and continue throughout the study period and for 90 days after the final study drug administration.
* Male subject must not donate sperm starting at Screening and throughout the study period and for 90 days after the final study drug administration.
* Subject has a Body Mass Index (BMI) range of 18.5 - 34.0 kg/m2 inclusive. The subject weighs at least 50 kg [at Screening].

Inclusion Criteria:Subjects with severe hepatic impairment must also meet the following inclusion criteria:

* Subject has a Child-Pugh classification Class C (severe, 10 to 15 points).

Inclusion Criteria: For Healthy Subjects Only:

* Age- and BMI-matched to subjects with severe liver hepatic impairment.

Exclusion Criteria:

* Subject has known or suspected hypersensitivity to enzalutamide, or any components of the formulation used.
* Subject has history of seizure or any condition that may predispose to seizure. Also history of loss of consciousness or transient ischemic attack within 12 months of enrollment (Day 1 visit).
* Subject has used grapefruit (or grapefruit containing products) or marmalade in the week prior to admission to the clinical unit (Day -1), as reported by the subject.

Exclusion Criteria: For Healthy Subjects Only:

* Subject has any of the liver function tests above the upper limit of normal.

Exclusion Criteria: Subjects with severe hepatic impairment must also not have any of the following characteristics:

* Subject has fluctuating or rapidly deteriorating hepatic function, as indicated by strongly varying or worsening of clinical and/or laboratory signs of hepatic impairment within the screening period.
* Subject has surgical porto-systemic shunts, including TIPSS (Trans-jugular intrahepatic portosystemic shunt).
* Subject has presence of severe hepatic encephalopathy (grade > 2).
* Subject has advanced ascites.
* Subject has esophageal variceal bleeding in the medical history (within 6 months before Day -1).
* Subject has thrombocyte level below 40x109 /L and /or hemoglobin below 90 g/L.
* Subject has significant renal dysfunction (creatinine clearance below 50 mL/min, estimated according to the method of Modification of Diet in Renal Disease (MDRD) formula).
* Subject has had previous liver transplantation.

Ages: 18 Years to 69 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of enzalutamide after a single oral dose | Days 1-6, 8, 12, 15, 19, 22, 26, 29, 36, 43, 50
  area under the plasma concentration - time curve (AUC) extrapolated to infinity (AUC0-inf)
PK of enzalutamide after a single oral dose | Days 1-6, 8, 12, 15, 19, 22, 26, 29, 36, 43, 50
  maximum concentration (observed) (Cmax)
PK of enzalutamide plus N-desmethyl enzalutamide (M2) after a single oral dose | Days 1-6, 8, 12, 15, 19, 22, 26, 29, 36, 43, 50
  area under the plasma concentration - time curve (AUC) extrapolated to infinity (AUC0-inf)
PK of enzalutamide plus N-desmethyl enzalutamide (M2) after a single oral dose | Days 1-6, 8, 12, 15, 19, 22, 26, 29, 36, 43, 50
  maximum concentration (observed) (Cmax)

SECONDARY OUTCOMES:
PK of enzalutamide, M1, M2 and the sum of enzalutamide plus N-desmethyl enzalutamide (M2) | Days 1-6, 8, 12, 15, 19, 22, 26, 29, 36, 43, 50
  Cmax and AUC0-inf (M1, M2 only), time to attain Cmax (tmax), AUC up to last quantifiable concentration (AUC0-last), apparent terminal elimination half life (t1/2), apparent volume of distribution during the terminal phase after extra vascular dosing (Vz/F), apparent total body clearance after extra vascular dosing (CL/F) (parent compound only), Metabolite-to-Parent Ratio (MPR), percent extrapolated for AUC0-inf (%AUC)
Additional pharmacokinetic variables for enzalutamide, and, as appropriate, for M1 and M2, based upon unbound plasma concentrations | Days 1-6, 8, 12, 15, 19, 22, 26, 29, 36, 43, 50
  Unbound Cmax (Cmax,u), unbound AUC0-inf (AUC0-inf,u), and unbound AUC0-last (AUC0-last,u). Unbound CL/F (CLu/F) and unbound Vz/F (Vz,u/F) (parent only)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Europe B.V.
Locations (1):
- Comac Medical Ltd., Sofia, Bulgaria